CLINICAL TRIAL: NCT04436484
Title: Immune Dysfunction in COVID-19: Investigation of Mechanisms and Identification of Immune Biomarkers of Clinical Outcome
Brief Title: Immune Biomarkers of Outcome From COVID-19
Acronym: IBOC
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20/HEP/381
Record Dates: First submitted 2020-06-12; First posted 2020-06-18 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: inflammation; immune response; biomarker
MeSH Terms: conditions — COVID-19; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Peripheral blood sampling — Non-interventional study

SUMMARY:
A new virus to humans, first identified in December 2019, is causing a global pandemic with over 1 million infections and many thousands of deaths. The virus, SARS-CoV2, leads to coronavirus disease 2019 (COVID-19), which mainly affects the breathing system. Around 1 in every 5 people with COVID-19 have more severe infection needing treatment in hospital. Up to half of them require help with breathing in an intensive care unit. Information we have so far about COVID-19 suggests that people with underlying conditions, such as high blood pressure and heart disease, or older people are at higher risk of having severe illness. Scientists do not yet understand why but think it may be related to the immune system.

SARS-CoV2 activates the immune system causing inflammation in the lungs, which is also seen in circulating immune cells in the blood. Preliminary reports show that the response of the immune system can be inappropriate, both overactive and also poorly responsive (exhausted). Changes in the type and function of immune cells have been linked to increased risk of severe disease or death from COVID-19.

In this study, the investigators will look for markers of immune function when a person first attends hospital, which can be used to predict whether they will go on to have a more severe infection. This will help treat patients more effectively, for example, by moving high risk patients to an intensive care setting at an early stage. The team will investigate the immune system in detail in 200 patients with COVID-19 attending University Hospitals Plymouth. The investigators will look for changes in the number, type and function of circulating immune cells and measure whether these changes are linked to severity of the infection or death. The investigators will use established techniques to measure immune function that could be rapidly put into routine hospital care to help guide treatment for individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending UHP with COVID-19 infection
* Participants capable of giving informed consent, or if not capable, assent from a personal or nominated consultee
* Age of 18 or over
* Confirmed COVID-19 infection by PCR or antibody testing

Exclusion Criteria:

* Participants on immune suppressing medications within preceding 4 weeks (including systemic corticosteroids with average daily dose equivalent to prednisolone 20 mg)
* Participants on treatment with systemic chemotherapy
* Participants with known immunodeficiency states
* Participants already administered immunomodulating or antiviral agents as part of an interventional trial (this does not include non-specific therapies such as hydroxycholoroquine)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with confirmed COVID-19 infection who are inpatients
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Mortality | up to 28 days
  Mortality

SECONDARY OUTCOMES:
Mortality | Day 4 and Day 10
  Mortality
Disease severity | Day 4, 10 and 28
  Sequential Organ Failure Assessment (SOFA) score (range 0-24; higher score predicts worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin D Dhanda, MRCP PhD, Principal Investigator — University Hospitals Plymouth NHS Trust
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Study findings will be reported but IPD is not planned to be shared.